CLINICAL TRIAL: NCT06820008
Title: Measurement and Impact of Physical Impairment in Amyotrophic Lateral Sclerosis: Use of Digital Technologies - A Precision ALS Project
Acronym: TechnicALS
Status: Recruiting | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Dara Meldrum, Associate Professor, Academic Unit of Neurology, Trinity College Dublin, University of Dublin, Trinity College
Other Study IDs: REC REF:24/17; Ref:240907 (Other: Trinity College Dublin Faculty of Heath Sciences Research Ethics Committee)
Record Dates: First submitted 2025-01-15; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neurone Disease
Keywords: ALS; PrecisionALS; Digital technologies; speech; swallow; dexterity; mobility; respiration; remote measurement; MND; outcome measurement
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Speech; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosed with the Amyotrophic Lateral Sclerosis (ALS) form of Motor Neurone Disease (MND).

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS), the most common form of Motor Neuron Disease (MND), is a neurodegenerative disease. At present there are limited treatment options for this disease which progressively affects physical function, i.e., the ability to speak, breathe, walk, and perform activities of daily living. ALS is a rare disease, and can present differently amongst individuals, therefore global collaboration is vital to have enough participants in studies to evaluate the effects of new treatments more precisely.

There are now many novel technologies that measure physical function which could be used in research studies to allow people with ALS to participate, in-part from home, knowing that they have access to the best clinical trials but with minimal time and travel burden. Their accuracy and the ability/willingness of people with ALS to use them need to be evaluated before they are accepted.

One of the traditional measurements used in research is called the ALS Functional Rating Scale -revised (ALSFRS-r) but this measurement has been criticised for being unable to pick up small changes and, in the digital age, outdated. The primary aim of this study is to develop a digital toolkit for more accurate measurement of physical aspects of ALS. It will test new technologies that measure physical function (i.e., walking, speech, swallow, strength, respiration (breathing), dexterity) that can be used by people with ALS in their own home.

This study has two aims:

Firstly, to test a selection of new digital technologies (in the form of devices, online systems and applications used on smartphones/electronic tablets) that measure physical function (e.g., walking, speech, strength) and assess whether the technologies are easy to use and acceptable both to people with ALS/MND and healthcare professionals.

Secondly, to measure how good technologies are at picking up changes in physical function over time and how they compare to older measures that are usually employed by clinicians.

This study will recruit 60 people with the ALS form of MND who attend a MND clinic in Dublin, Ireland. The study will run from November 2024 to December 2027 approximately. During this period, each participant will be asked to take part for a duration of 12 months.

The study will compare measurements of physical function collected by a researcher in the traditional way, with new ways of measuring the same functions, using technologies that can be used at home by the person with ALS. The experience of people using the technologies at home will be evaluated with interviews and questionnaires.

Over the 12-month duration, participants will be assessed in person by members of the research team on 3 occasions. These assessments will be carried out in the clinic setting or can be completed at the participant's home instead if needed.

In between the in-person assessments, participants will also do assessments in their own home every week using technologies, either independently or with telephone or video support from a researcher. The technologies that the participant use at home will be matched to the ones that were assigned to them for the in-person assessment at the beginning. Participants will use only technologies that are suited to them. The researcher will talk to participants about which technologies are suitable for them and which they are comfortable to use.

Participants coded data collected using the new technologies will be analyzed using established methods and newer methods such as artificial intelligence (AI). AI refers to the ability of computers and digital devices to learn and simulate human intelligence. Machine learning, a field within AI, analyses large data sets to develop models that improve as more data is added. Analysis of participants coded data will be for research purposes only and will not be used for their medical care.

Ultimately this study will create new knowledge on the role of technology in physical measurement in MND and how it can be successfully used in future studies to help find effective treatments.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the validity and usability of novel digital technologies in the measurement of physical impairments (speech, swallow, strength, dexterity, mobility, and respiration) in ALS and the adherence to their use over time. The technologies that will be used in the study are as follows:

1. Speech Intelligibility Test (SIT) - software that measures speech intelligibility
2. ModalityAi- an online system that collects and analyses speech samples
3. Iowa Oral Performance Instrument (IOPI) - a device that measures tongue strength and endurance
4. Grip dynamometer - a device that measures grip strength
5. Index-eTap - a novel device and an app that measure dexterity
6. GaitKeeper - an app that measures walking
7. ActiGraph - a device that measures physical activity
8. MIR Spirometer - a device and app that measure breathing
9. Telehealth in Motor Neurone Disease (TiM) - an app that measures symptoms reported by the participant (patient reported outcome measures)

Usability will be measured by means of a questionnaire called the System Usability Scale (SUS) and a semi-structured interview with a researcher.

The objectives of the study are to:

1. Quantify the adherence to, usability and validity of novel digital technologies in measurement of physical parameters in ALS.
2. To compare the adherence to, usability and validity of actigraphy with devices worn on the wrist and hip concurrently for remote activity measurement.
3. To compare the adherence to, usability and validity of remote spirometry conducted independently or with clinician support via video consultation.
4. To examine the ability of Index-eTap to detect meaningful change over time in people with ALS/MND.
5. To examine the impact of impairments in cognition and behaviour on the use of digital technologies.
6. To examine the utility of audio-visual recordings for multimodal analysis of speaker samples using Modality software to analyse speech, cognitive-linguistic and facial muscle movement metrics.
7. To investigate the validity of combining data from validated technologies to form a unified scale sensitive to changes in physical impairments in ALS.
8. To develop optimal methods of summarising and visualising data relating to ALS physical impairments, for researchers working in the field of ALS

Participants will complete regular assessments of physical function remotely ('at-home') using novel digital technologies and will in parallel complete three researcher-led ('in-person') assessments of comparable constructs. The in-person assessments will take place either in the clinical research centre, Beaumont Hospital or during an outreach home visit by a member of the research team, based on participant preference. On recruitment to the study, baseline demographic and clinical information will be collected from the participant and their Beaumont Hospital medical record. Participants will be followed up for one year. Participants will be recruited over 18 months. The anticipated total study duration is approximately 3 years, including data analysis.

In-person assessments: The researcher will administer traditional assessments (as gold standard comparison for remote measurements) and will complete assessments using novel technologies where appropriate. In-person assessments will take place at baseline, 3 months and 12 months (or at withdrawal from the study).

This assessment battery will include:

* Speech intelligibility/rate: assessed using Speech Intelligibility Test (SIT) software and Zoom H1 dictaphone (traditional assessment)
* Tongue strength and endurance: assessed using Iowa Oral Performance Instrument (IOPI) Pro device (traditional assessment)
* Hand grip strength: Analogue Jamar Hydraulic Handgrip Dynamometer (traditional assessment)
* Finger dexterity: Index-eTap device (this is a prototype device which is currently only suitable for use with a researcher and will be completed in person)
* Mobility: GaitKeeper (this is a research-use novel gait analysis system, which requires testing in ALS for both in-person and for remote use)
* Slow Vital Capacity (SVC): assessed using Micro Medical or equivalent desktop Spirometer device (traditional assessment)
* Sniff Nasal Inspiratory Pressure (SNIP): assessed using MicroRPM device (traditional assessment)
* Peak Cough Flow (PCF): Analogue peak flow meter device and facemask (traditional assessment)

Additionally traditional validated questionnaires and rating scales will be completed:

* Bulbar function: Centre for Neurological Studies Bulbar Function Scale (CNS-BFS)
* Food texture description: Functional Oral Intake Scale (FOIS)
* Upper limb function: Disability of Arm, Shoulder and Hand (DASH)
* Overall function: ALS Functional Rating Scale - revised (ALSFRS-r)

Following the baseline assessments, participants will be provided with the technologies appropriate for their use at home and will be trained in their use. Thereafter, participants will complete 'at-home' assessments, using technologies either independently or with support via video or phone call following a defined schedule. Participants will be asked to use a minimum of 2 suitable technologies, which will be selected by the researchers based on their clinical presentation. Participants will be provided with the option to opt-out of using a technology that they feel it would be overly burdensome for them. Researchers will maintain regular contact with participants, via phone call or video call and will 'check-in' regularly regarding how they are managing with the at-home assessments.

These will include:

* Multimodal assessment of speech and facial movement: using the Modality online system
* Tongue strength: using Iowa Oral Performance Instrument (IOPI) Trainer device
* Hand grip strength: Prototype strength ergometer device (5 participants will use this novel prototype device designed in Trinity College Dublin)
* Mobility: using GaitKeeper app
* Activity: using ActiGraph GT9X Link device to monitor activity
* Slow Vital Capacity (SVC): using Medical International Research (MIR) Spirobank Smart spirometer device. This is used with an app and will be completed every second month via video call and every second month independently by the participant guided by the app.
* Peak Cough Flow (PCF): using an analogue peak flow meter device (completed independently with score entered on TiM).
* Telehealth in MND (TiM) on MyPathway: a remote monitoring system where patient-reported outcome measures are completed online. This is currently in clinical use in the Beaumont Hospital clinical service. It will collect usual questionnaires and study specific questionnaires
* Communication Effectiveness Index - modified (CETI-m)
* Eating Assessment Tool (EAT-10)
* ALSFRS-r (self-reported)

Validity of the remote measures and the novel technologies will be assessed by comparing traditional assessment methods to novel methods. After using a technology at least twice, a subset of participants will be invited to complete the System Usability Scale (SUS) questionnaire and a semi-structured interview regarding their experience using the technology. Percentage adherence to the remote monitoring schedule will also be quantified. The study will operate in accordance with data protection legislation (GDPR), the declaration of Helsinki, and with Irish and EU legal and ethical requirement for cyber-protection of sensitive patient data. A data protection impact assessment (DPIA) has been completed and approved by the Beaumont Hospital and Trinity College Dublin ethics boards. Data sharing agreements are also in place for any of the relevant technologies included in the study.

This study is part of a larger research program entitled Precision ALS [www.precisionals.ie]. Precision ALS is a European project which aims to collect large amounts of data about people with MND all over Europe, to make research in ALS/MND more powerful.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS made by a Neurologist; possible, lab-supported probable, probable or definite as per the revised El Escorial Criteria.
* Enrolled in the Precision ALS prospective study.
* Ability to understand participation requirements and provide informed consent to undergo assessments and for data to be used.
* Willingness to use a smartphone or tablet and to download and use study apps.
* Age >18 years
* Home access to a stable broadband internet connection and willingness to use this for data collection.

Exclusion Criteria:

* Diagnosis of a neurological disease other than ALS, active dementia or psychiatric illness that would limit ability to follow the assessment schedule of the study.
* Other medical condition that would compromise the patient's safety or limit their participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will primarily take place at the MND clinic in a hospital in Dublin, Ireland (Beaumont Hospital). The national support organisation, the Irish Motor Neurone Disease Association (IMNDA), will also share information about the study including contact details for the research team to their clients through their website and quarterly member's newsletter.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Completion of 12-month follow up period | 12 months per participant
  An adherence percentage will be calculated based on the number of data captures completed by the participant divided by the total target number of data captures multiplied by 100/1.
System Usability Scale | Modality (Month 1), IOPI Trainer (Month 5), Prototype hand grip ergometer (after 2/3 uses), Index-eTap (Month 3), GaitKeeper (Month 3), ActiGraph (Month 3), MIR (Month 5), PCF (Month 3)
  A system usability scale (SUS) will be carried out on every technology to assess usability with a sample of 15 patients per technology (except the prototype hand grip ergometer which will have a sample of 5 patients). Responses will be collected once for each remote or prototype technology that the participant uses over the course of the study. The participant will have used the technology at least twice prior to collecting feedback and as such this affects the schedule for the SUS interviews. Technologies that are part of the in-person assessments (Index-eTap and Gaitkeeper) will have their SUS interviews scheduled in Month 3 (second in-person visit). All other technologies will have their SUS interviews carried out at least 2/3 uses via a video call and before 5 months. This is to reduce burden on participants.

SECONDARY OUTCOMES:
Participant withdrawal or death during the study. | Less than 12 months depending on date of participant withdrawal or death.
  Date of withdrawal or death will be recorded. A percentage attrition rate will be calculated based on the number of participants who withdrew or died within the 12-month period divided by the total number of participants who completed baseline functional measures multiplied by 100/1
Semi-structured interview on usability | Modality (Month 1), IOPI Trainer (Month 5), Prototype hand grip ergometer (after 2/3 uses), Index-eTap (Month 3), GaitKeeper (Month 3), ActiGraph (Month 3), MIR (Month 5), PCF (Month 3)
  Semi-structured interviews on usability will be carried out on every technology to assess usability with a sample of 15 patients per technology (except the prototype hand grip ergometer which will have a sample of 5 patients). Responses will be collected once for each remote or prototype technology that the participant uses over the course of the study. The participant will have used the technology at least twice prior to collecting feedback and as such this affects the schedule for the interviews. Technologies that are part of the in-person assessments (Index-eTap and Gaitkeeper) will have their interviews scheduled in Month 3 (second in-person visit). All other technologies will have their interviews carried out at least 2/3 uses via a video call and before 5 months. This is to reduce burden on participants.

CONTACTS AND LOCATIONS:
Overall Officials: Dara Meldrum, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Beaumont Hospital, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Data will only be analysed by researchers within the Precision ALS partnership within their host institutions in coordination with the local and overall PIs. Data analysis permissions are also governed by the inter-institutional agreement.